CLINICAL TRIAL: NCT01109004
Title: A Trial of Single Autologous Transplant With or Without Consolidation Therapy Versus Tandem Autologous Transplant With Lenalidomide Maintenance for Patients With Multiple Myeloma (BMT CTN 0702)
Brief Title: Stem Cell Transplant With Lenalidomide Maintenance in Patients With Multiple Myeloma (BMT CTN 0702)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0702; BMT CTN 0702 (Other: Blood and Marrow Transplant Clinicial Trials Network); U01HL069294-05 (NIH); 690 (Other: National Heart, Lung, and Blood Institute); NCT02257515 (obsolete NCT alias)
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma
Keywords: Symptomatic Multiple Myeloma; Lenalidomide; Anti-Myeloma Agents; Hematologic Disorders; Maintenance Therapy; Progression; Autologous Transplant; RVD Consolidation
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases; Disease Progression | interventions — Lenalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tandem auto transplant (Active Comparator): Initial autologous transplant followed by a second autologous transplant and lenalidomide maintenance
  Interventions: Drug: Lenalidomide
- RVD consolidation (Active Comparator): Initial autologous transplant followed by lenalidomide, bortezomib and dexamethasone (RVD) consolidation and lenalidomide maintenance
  Interventions: Drug: lenalidomide, bortezomib and dexamethasone
- Lenalidomide maintenance (Active Comparator): Initial autologous transplant followed by lenalidomide maintenance
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — All patients will undergo a first autologous peripheral blood stem cell (PBSC) transplant with high-dose melphalan (200 mg/m^2 IV) given on Day -2. Upon recovery from the first transplant patients will receive a second autologous PBSC transplant with the same conditioning regimen as the first transplant. All patients will also receive maintenance lenalidomide which will start after the second transplant. Maintenance therapy with lenalidomide will start at 10 mg daily for 3 months and increase to 15 mg daily. The duration of maintenance will be three years in all treatment arms.
  Other Names: Revlimid™
  Arms: Tandem auto transplant
Drug: lenalidomide, bortezomib and dexamethasone — All patients will undergo a first autologous peripheral blood stem cell (PBSC) transplant with high-dose melphalan (200 mg/m^2 IV) given on Day -2. Upon recovery from the first transplant patients will receive consolidation therapy with RVD (lenalidomide 15 mg/day on Days 1-14, dexamethasone 40mg on Days 1, 8 and 15, and bortezomib 1.3mg/m2 on Days 1, 4, 8 and 11 of every 21 day cycle, patients will receive four cycles). All patients will also receive maintenance lenalidomide which will start after consolidation therapy. Maintenance therapy with lenalidomide will start at 10 mg daily for 3 months and increase to 15 mg daily. The duration of maintenance will be three years in all treatment arms.
  Other Names: Revlimid™, Velcade®, and Decadron
  Arms: RVD consolidation
Drug: Lenalidomide — All patients will undergo a first autologous peripheral blood stem cell (PBSC) transplant with high-dose melphalan (200 mg/m^2 IV) given on Day -2. Upon recovery from the first transplant patients will receive maintenance with lenalidomide (15 mg daily). Maintenance lenalidomide will start after the first autologous transplant. Maintenance therapy with lenalidomide will start at 10 mg daily for 3 months and increase to 15 mg daily. The duration of maintenance will be three years in all treatment arms.
  Other Names: Revlimid™
  Arms: Lenalidomide maintenance

SUMMARY:
The study is designed as a Phase III, multicenter trial of tandem autologous transplants plus maintenance therapy versus the strategy of single autologous transplant plus consolidation therapy with lenalidomide, bortezomib and dexamethasone (RVD) followed by maintenance therapy or single autologous transplant plus maintenance therapy as part of upfront treatment of multiple myeloma (MM). Lenalidomide will be used as maintenance therapy for three years in all arms.

DETAILED DESCRIPTION:
The primary objective of the randomized trial is to compare three-year progression-free survival (PFS) between the three treatment arms as a pairwise comparison. Mobilization therapy will not be specified for the study. Randomization to three treatment arms will be done prior to the first transplants. All patients will undergo a first autologous peripheral blood stem cell (PBSC) transplant with high-dose melphalan (200 mg/m^2 IV) given on Day -2. Upon recovery from the first transplant patients will receive either a second autologous PBSC transplant with the same conditioning regimen as the first transplant or consolidation therapy with RVD (lenalidomide 15 mg/day on Days 1-14, dexamethasone 40 mg on Days 1, 8 and 15, and bortezomib 1.3mg/m^2 on Days 1, 4, 8 and 11 of every 21 day cycle, patients will receive four cycles) or maintenance with lenalidomide (15 mg daily). All patients will also receive maintenance lenalidomide which will start after the second transplant, after the first autologous transplant or after consolidation therapy depending on the treatment arm. Maintenance therapy with lenalidomide will start at 10 mg daily for three months and increase to 15 mg daily. The duration of maintenance will be three years in all treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the criteria for symptomatic multiple myeloma (MM).
* Patients who are 70 years of age, or younger, at time of enrollment.
* Patients who have received at least two cycles of any regimen as initial systemic therapy and are within 2 - 12 months of the first dose of initial therapy.
* Cardiac function: left ventricular ejection fraction at rest greater than 40 percent.
* Hepatic: bilirubin less than 1.5x the upper limit of normal and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 2.5x the upper limit of normal. (Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value of 1.5x the upper limit of normal.)
* Renal: Creatinine clearance of grater than or equal to 40 mL/min, estimated or calculated.
* Pulmonary: Diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) greater than 50 percent of predicted value (corrected for hemoglobin).
* Patients with an adequate autologous graft defined as a cryopreserved PBSC graft containing greater than or equal to 4 x 10^6 CD34+ cells/kg patient weight. The graft may not be CD34+ selected or otherwise manipulated to remove tumor or other cells. The graft can be collected at the transplanting institution or by a referring center. The autograft must be stored so that there are two products each containing at least 2 x 10^6 CD34+ cells/kg patient weight.
* Signed informed consent form.

Exclusion Criteria:

* Patients who never fulfill the criteria for symptomatic MM.
* Patients with purely non-secretory MM [absence of a monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques]. Patients with light chain MM detected in the serum by free light chain assay are eligible.
* Patients with plasma cell leukemia.
* Karnofsky performance score less than 70 percent.
* Patients with greater than grade 2 sensory neuropathy (CTCAE).
* Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms).
* Patients seropositive for the human immunodeficiency virus (HIV).
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received other investigational drugs with 14 days before enrollment.
* Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs. Cancer treated with curative intent greater than 5 years previously is allowed.
* Female patients who are pregnant (positive B-HCG) or breastfeeding.
* Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use contraceptive techniques during the length of lenalidomide maintenance therapy.
* Prior allograft or prior autograft.
* Patients who have received mid-intensity melphalan (greater than 50 mg IV) as part of prior therapy.
* Patients unable or unwilling to provide informed consent.
* Prior organ transplant requiring immunosuppressive therapy.
* Patients with disease progression prior to enrollment.
* Patients who have received lenalidomide as initial therapy for MM and have experienced toxicities resulting in treatment discontinuation.
* Patients who experienced thromboembolic events while on full anticoagulation during prior therapy with lenalidomide or thalidomide.
* Patients unwilling to take deep vein thrombosis (DVT) prophylaxis.
* Patients who cannot undergo an intervention in any treatment arm due to a priori denial of medical costs coverage by third party payers.
* Patients unable to unwilling to return to the transplant center for their assigned treatments.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (54):
- United States (54):
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UCSD Medical Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Christiana Care Health System, Newark, Delaware
  - University of Florida College of Medicine, Gainesville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Blood and Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - St. Lukes Mountain States Tumor Institute, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Wichita CCOP, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - DFCI, Brigham and Womens Hospital, Boston, Massachusetts
  - DFCI, Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - North Shore University Hospital, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State College of Medicine, The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Sarah Cannon Blood & Marrow Transplant Program, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas, MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Stadtmauer EA, Pasquini MC, Blackwell B, Hari P, Bashey A, Devine S, Efebera Y, Ganguly S, Gasparetto C, Geller N, Horowitz MM, Koreth J, Knust K, Landau H, Brunstein C, McCarthy P, Nelson C, Qazilbash MH, Shah N, Vesole DH, Vij R, Vogl DT, Giralt S, Somlo G, Krishnan A. Autologous Transplantation, Consolidation, and Maintenance Therapy in Multiple Myeloma: Results of the BMT CTN 0702 Trial. J Clin Oncol. 2019 Mar 1;37(7):589-597. doi: 10.1200/JCO.18.00685. Epub 2019 Jan 17. PMID 30653422
- [Derived] Pasquini MC, Wallace PK, Logan B, Kaur M, Tario JD, Howard A, Zhang Y, Brunstein C, Efebera Y, Geller N, Giralt S, Hari P, Horowitz MM, Koreth J, Krishnan A, Landau H, Somlo G, Shah N, Stadtmauer E, Vogl DT, Vesole DH, McCarthy PL, Hahn T. Minimal Residual Disease Status in Multiple Myeloma 1 Year After Autologous Hematopoietic Cell Transplantation and Lenalidomide Maintenance Are Associated With Long-Term Overall Survival. J Clin Oncol. 2024 Aug 10;42(23):2757-2768. doi: 10.1200/JCO.23.00934. Epub 2024 May 3. PMID 38701390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Started | 247 | 254 | 257
Completed | 247 | 254 | 257
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance | Total
Number analyzed (Participants) | 247 | 254 | 257 | 758
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 70] | 57 [20 to 70] | 56 [30 to 70] | 56 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 108 | 96 | 304
  Male | 147 | 146 | 161 | 454
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 178 | 192 | 201 | 571
  African American | 50 | 39 | 41 | 130
  Multiple/Other/Unknown | 19 | 23 | 15 | 57
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    90 or Greater | 182 | 169 | 172 | 523
    Less Than 90 | 65 | 85 | 85 | 235
Disease Risk [Count of Participants; unit: Participants] — Participants on this study will be stratified for the purposes of statistical analysis into high-risk and standard risk-groups. High-risk multiple myeloma is defined by the presence of high beta-2 microglobulin (> 5.5mg/L) or the presence of cytogenetic abnormalities including t(4;14), t(14;20), t(14;16), deletion (17p) detected by FISH or standard cytogenetics, deletion 13 detected by standard cytogenetics only or aneuploidy. Participants without cytogenetic analysis available and beta-2 microglobulin ≤ 5.5mg/L or with deletion 13 detected by FISH will be classified as standard-risk disease.
  Participants
    Standard | 175 | 178 | 182 | 535
    High | 72 | 76 | 75 | 223
Initial Therapy [Count of Participants; unit: Participants] — Initial therapy administered for the treatment of multiple myeloma
  Participants
    Bortezomib/Lenalidomide/Dexamethasone | 141 | 136 | 143 | 420
    Bortezomib/Cyclophosphamide/Dexamethasone | 33 | 35 | 40 | 108
    Lenalidomide/Dexamethasone | 24 | 28 | 22 | 74
    Bortezomib/Dexamethasone | 29 | 32 | 32 | 93
    Other | 19 | 19 | 20 | 58
    Unknown | 1 | 4 | 0 | 5
Time from Initial Therapy to Enrollment [Median (Full Range); unit: months] | 5 [2 to 14] | 5 [2 to 12] | 5 [2 to 12] | 5 [2 to 14]
Number of Lines of Therapy [Count of Participants; unit: Participants] — Lines of therapy is defined as the number of different regimens received prior to study entry.
  Participants
    1 | 210 | 213 | 218 | 641
    2 | 31 | 36 | 37 | 104
    3 | 5 | 1 | 2 | 8
    Unknown | 1 | 4 | 0 | 5
Disease Status at Enrollment [Count of Participants; unit: Participants]
  Stringent Complete Response | 21 | 26 | 23 | 70
  Complete Response | 22 | 19 | 24 | 65
  Near Complete Response | 27 | 22 | 24 | 73
  Very Good Partial Response | 52 | 53 | 43 | 148
  Partial Response | 106 | 108 | 123 | 337
  Stable Disease | 14 | 21 | 14 | 49
  Progression | 4 | 2 | 3 | 9
  Not Evaluable | 1 | 3 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: Progression-free survival is defined as survival without disease progression or initiation of non-protocol anti-myeloma therapy. To account for loss to follow-up of a few participants, the Kaplan-Meier estimator was used to estimate progression-free survival at 38 months post-randomization.
Time Frame: 38 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 58.5 [51.7 to 64.6] | 57.8 [51.4 to 63.7] | 53.9 [47.4 to 60.0]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with PFS at 38 months post-randomization are equal for those receiving Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.87, Log Rank — The primary analysis involved pairwise comparisons of PFS between the three treatment arms. To control the familywise type I error rate at 0.05, two-sided testing was performed at a Bonferroni-adjusted significance level of 0.0167 = 0.05 / 3; The log rank test was stratified on risk status (high risk vs. standard risk)
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with PFS at 38 months post-randomization are equal for those receiving Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.37, Log Rank — [p-value comment as in outcome 1, analysis 1]; The log rank test was stratified on risk status (high risk vs. standard risk)
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with PFS at 38 months post-randomization are equal for those receiving RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.27, Log Rank — [p-value comment as in outcome 1, analysis 1]; The log rank test was stratified on risk status (high risk vs. standard risk)

2. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease Progression is defined as progression of multiple myeloma, including one or more of the following:
  * A reappearance of serum monoclonal paraprotein, with a level of at least 0.5 g/dL
  * 24-hour urine protein electrophoresis with at least 200 mg paraprotein/24 hours
  * Abnormal free light chain levels of >10 mg/dl, only in patients without measurable paraprotein in the serum and urine
  * At least 10% plasma cells in a bone marrow aspirate or on trephine biopsy
  * Definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of new bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia (corrected serum Ca >11.5 mg/dL or >2.8 mmol/L) not attributable to any other cause
  To account for loss to follow-up of a few participants, the cumulative incidence of TRM at 38 months post-randomization was estimated using the Aalen-Johansen estimator, treating death prior to disease progression as a competing risk.
Time Frame: 38 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 39.8 [33.4 to 46.1] | 41.0 [34.7 to 47.0] | 45.6 [39.2 to 51.8]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with disease progression at 38 months post-randomization are equal for those receiving Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.92, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with disease progression at 38 months post-randomization are equal for those receiving Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.21, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with disease progression at 38 months post-randomization are equal for those receiving RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.22, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk

3. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival is defined as survival of death from any cause. To account for loss to follow-up of a few participants, the Kaplan-Meier estimator was used to estimate overall survival at 38 months post-randomization.
Time Frame: 38 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 81.8 [76.2 to 86.2] | 85.4 [80.4 to 89.3] | 83.7 [78.4 to 87.8]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with OS at 38 months post-randomization are equal for those receiving Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.26, Log Rank — Two sided testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with OS at 38 months post-randomization are equal for those receiving Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.53, Log Rank — Two sided testing was performed at a significance level of 0.05
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with OS at 38 months post-randomization are equal for those receiving RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.57, Log Rank — Two sided testing was performed at a significance level of 0.05

4. Secondary Outcome: Percentage of Participants With Treatment-related Mortality (TRM)
Description: TRM is defined as death prior to progression of multiple myeloma. To account for loss to follow-up of a few participants, the cumulative incidence of TRM at 38 months post-randomization was estimated using the Aalen-Johansen estimator, treating disease progression as a competing risk.
Time Frame: Up to 38 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 1.7 [0.6 to 4.2] | 1.2 [0.3 to 3.3] | 0.5 [0.0 to 2.4]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with TRM at 38 months post-randomization are equal for those receiving Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.63, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with TRM at 38 months post-randomization are equal for those receiving Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.15, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with TRM at 38 months post-randomization are equal for those receiving RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.33, Gray's test — Two sided testing was performed at a significance level of 0.05; Death prior to disease progression was treated as a competing risk

5. Secondary Outcome: Number of Participants With Treatment Response
Description: The number of participants with very good partial response (VGPR) or better [complete response (CR), near CR (nCR), and stringent CR (sCR)] according to the International Uniform Response Criteria will be calculated. The "Worse than VGPR" group includes PR, stable disease, and progressive disease.
  sCR requires, in addition to CR: Normal free light chain ratio (FLC), Absence of clonal cells in bone marrow CR requires, in addition to nCR: Absence of the original monoclonal paraprotein (PPN), Disappearance of soft tissue plasmacytomas nCR is defined as: < 5% plasma cells in a bone marrow aspirate, No increase in lytic bone lesions VGPR requires: Serum or urine PPN not detectable on electrophoresis OR >=90% reduction in serum PPN plus urine PPN <100 mg/24hrs, >= 50% reduction in the level of serum monoclonal PPN or reduction in 24 hour urinary monoclonal PPN either >= 90% or to <200 mg/24 hours in light chain disease, >= 50% reduction in the size of soft tissue plasmacytomas
Time Frame: 1 and 2 years post-randomization
Population: Only participants that were evaluable for disease response were analyzed at each time point. Those who had died or experienced disease progression were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
Participants
  1 Year: number analyzed (Participants) | 192 | 209 | 208
  1 Year: CR or sCR | 97 | 122 | 98
  1 Year: VGPR or nCR | 56 | 50 | 60
  1 Year: Worse than VGPR | 39 | 37 | 50
  2 Years: number analyzed (Participants) | 157 | 175 | 160
  2 Years: CR or sCR | 98 | 117 | 93
  2 Years: VGPR or nCR | 39 | 37 | 41
  2 Years: Worse than VGPR | 20 | 21 | 26

6. Secondary Outcome: FACT-G Total Score
Description: The Functional Assessment of Cancer Therapy-General (FACT-G) is a quality of life instrument that assesses the effects of cancer therapy on a patient's physical, social/family, emotional, and functional well-being. The assessment has 27 questions, each scored on a Likert scale from 0-4. The overall score is computed by adding scores of the questions and falls in the range 0-108, with higher scores indicating higher levels of overall well-being.
Time Frame: Up to 3 years post-randomization
Population: Outcomes are analyzed from participants that were alive, progression-free, and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
score on a scale
  Baseline: number analyzed (Participants) | 226 | 220 | 233
  Baseline | 79 (1.0) | 79 (1.0) | 77 (1.0)
  1 Year: number analyzed (Participants) | 162 | 172 | 177
  1 Year | 84 (1.3) | 84 (1.3) | 83 (1.2)
  2 Years: number analyzed (Participants) | 127 | 140 | 128
  2 Years | 84 (1.5) | 84 (1.3) | 85 (1.4)
  3 Years: number analyzed (Participants) | 98 | 107 | 96
  3 Years | 85 (1.6) | 84 (1.6) | 85 (1.7)

7. Secondary Outcome: FACT-BMT Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant scale (FACT-BMT) is a quality of life instrument that assesses the effects of bone marrow transplantation (BMT) on a patient's physical, social/family, emotional, and functional well-being while taking into consideration BMT-specific concerns. The assessment has 37 questions, each scored on a Likert scale from 0-4. The overall score is computed by adding scores of the questions and falls in the range 0-148, with higher scores indicating higher levels of overall well-being.
Time Frame: Up to 3 years post-randomization
Population: Outcomes are analyzed from participants that were alive, progression-free, and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
score on a scale
  Baseline: number analyzed (Participants) | 225 | 219 | 233
  Baseline | 107 (1.4) | 107 (1.3) | 105 (1.3)
  1 Year: number analyzed (Participants) | 162 | 172 | 177
  1 Year | 113 (1.7) | 115 (1.7) | 113 (1.6)
  2 Years: number analyzed (Participants) | 127 | 139 | 128
  2 Years | 114 (1.8) | 115 (1.7) | 115 (1.7)
  3 Years: number analyzed (Participants) | 98 | 107 | 96
  3 Years | 115 (2.0) | 114 (2.1) | 115 (2.2)

8. Secondary Outcome: FACT-BMT Trial Outcome Index
Description: The Functional Assessment of Cancer Therapy (FACT) Trial Outcome Index is a quality of life instrument that assesses the impact of bone marrow transplantation (BMT) on a patient's physical and functional well-being while taking into consideration BMT-specific concerns. The assessment has 24 questions, each scored on a Likert scale from 0-4. The overall score is computed by adding scores of the questions and falls in the range 0-96, with higher scores indicating higher levels of overall well-being.
Time Frame: Up to 3 years post-randomization
Population: Outcomes are analyzed from participants that were alive, progression-free, and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
score on a scale
  Baseline: number analyzed (Participants) | 226 | 220 | 233
  Baseline | 64 (1.1) | 65 (1.0) | 63 (1.0)
  1 Year: number analyzed (Participants) | 162 | 172 | 177
  1 Year | 70 (1.2) | 72 (1.2) | 71 (1.1)
  2 Years: number analyzed (Participants) | 126 | 139 | 128
  2 Years | 73 (1.2) | 73 (1.3) | 73 (1.2)
  3 Years: number analyzed (Participants) | 98 | 108 | 96
  3 Years | 73 (1.4) | 71 (1.5) | 73 (1.5)

9. Secondary Outcome: MOS SF-36 Physical Component Summary
Description: The Medical Outcome Study (MOS) SF-36 Physical Component Summary is a subscale of the SF-36 intended to measure physical well-being. It is scored on a scale of 0-100, with higher scores indicating higher levels of well-being.
Time Frame: Up to 3 years post-randomization
Population: Outcomes are analyzed from participants that were alive, progression-free, and completed assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
score on a scale
  Baseline: number analyzed (Participants) | 220 | 221 | 228
  Baseline | 37 (0.7) | 39 (0.7) | 38 (0.7)
  1 Year: number analyzed (Participants) | 159 | 166 | 176
  1 Year | 43 (0.8) | 43 (0.8) | 42 (0.7)
  2 Years: number analyzed (Participants) | 124 | 137 | 124
  2 Years | 44 (0.8) | 44 (0.9) | 43 (0.9)
  3 Years: number analyzed (Participants) | 94 | 107 | 95
  3 Years | 42 (1.0) | 42 (1.0) | 43 (1.0)

10. Secondary Outcome: MOS SF-36 Mental Component Summary
Description: The Medical Outcome Study (MOS) SF-36 Mental Component Summary is a subscale of the SF-36 intended to measure mental well-being. It is scored on a scale of 0-100, with higher scores indicating higher levels of well-being.
Time Frame: Up to 3 years post-randomization
Population: Outcomes are analyzed from participants that were alive, progression-free, and completed assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
score on a scale
  Baseline: number analyzed (Participants) | 220 | 221 | 228
  Baseline | 49 (0.7) | 48 (0.7) | 48 (0.8)
  1 Year: number analyzed (Participants) | 159 | 166 | 176
  1 Year | 50 (0.9) | 51 (0.8) | 50 (0.8)
  2 Years: number analyzed (Participants) | 124 | 137 | 124
  2 Years | 50 (1.0) | 50 (0.8) | 50 (1.0)
  3 Years: number analyzed (Participants) | 94 | 107 | 95
  3 Years | 51 (1.0) | 50 (1.1) | 51 (1.0)

ADVERSE EVENTS:
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Serious Adverse Events (participants affected / at risk) | 42/247 | 45/254 | 53/257
Other Adverse Events (participants affected / at risk) | 0/247 | 0/254 | 0/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Auto Transplant (N=247) | RVD Consolidation (N=254) | Lenalidomide Maintenance (N=257)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Arthroscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No